CLINICAL TRIAL: NCT06607315
Title: The Relationship Between Running Form, Soft Tissue Physical Properties, and Injury in Long-Distance Runners
Brief Title: Soft Tissue Physical Properties in Long-Distance Runners
Status: Not yet recruiting | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Okan University (Other)
Responsible Party: Principal Investigator, Gamze Aydin, Principal Investigator, Istanbul University - Cerrahpasa
Other Study IDs: IstanbulOkanUn
Record Dates: First submitted 2024-09-12; First posted 2024-09-23 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Runner
Keywords: soft tissue; injury; running
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: physical properties of soft tissue — Using the Myoton Pro device, the physical properties such as elasticity and viscosity of the Achilles tendon, patellar tendon, gastrocnemius, quadriceps, and hamstring muscles will be measured.
Other: Analysis of Running Form — High-speed camera systems will be used to analyze biomechanical parameters in detail, such as angular movements of the lower extremity joints (tibia, ankle, knee, hip), step length, and ground contact time during running. These analyses will allow us to objectively characterize different running forms.

SUMMARY:
The aim of this study is to investigate in greater depth the effects of different running forms on soft tissue physical properties in long-distance runners and the relationship of this to injury risk. By doing so, the study seeks to provide new insights into the pathophysiology of running injuries and develop more effective injury prevention strategies.

DETAILED DESCRIPTION:
This study is expected to reveal the effects of different running forms on soft tissue physical properties in long-distance runners and the relationship of these effects to injury risk.

Running analysis will be conducted by recording 30-second videos of participants during their runs, and tests will be performed using the MyotonePro device on predetermined areas. Before the evaluations, all participants will be informed about the study's objectives and their verbal informed consent will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* individuals who have been regularly running long distances for at least 1 year,
* between the ages of 25 and 35,
* classified as amateur athletes

Exclusion Criteria:

* Having undergone orthopedic surgery involving the lower extremity

Ages: 25 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: between the ages of 25 and 35 individuals who have been regularly running long distances for at least 1 year
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2024-12-15 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
myoton pro device | 3 months
  the physical properties of the tendon will be measure
running form analysis | 3 months
  High-speed camera systems will be used to analyze biomechanical parameter of lower extremity

CONTACTS AND LOCATIONS:
Locations (1):
- Gamze Aydın, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No